CLINICAL TRIAL: NCT06374836
Title: To Quantify the Contractile Response of the Thoracic Aorta to Vasoactive Substances and Identify Potential Predictors of This Response.
Brief Title: The Contractile Response of the Thoracic Aorta to Vasoactive Substances
Acronym: AorticContract
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Principal Investigator, Frederique de Raat, Principal investigator, Catharina Ziekenhuis Eindhoven
Other Study IDs: nWMO 2024.040
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-09

CONDITIONS: Human Thoracic Aorta Contractility
MeSH Terms: interventions — Phenylephrine; Nitroprusside; Nicardipine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Phenylephrine — At the OR, the patient will be sedated and have a transoesophageal echo (TEE) catether inserted, which is part of standard clinical care. When a patient becomes hypotensive and the attending anesthesiologist decides to infuse any of the following drugs (phenylephrine, ephedrine, norepinephrine, nitroprusside, or nicardipine), before infusion, the anesthesiolgist will acquire with TEE 10 beats of the thoracic ascending and descending aorta respectively. This is defined as one measurement. Five minutes after infusion the same measurement is repeated. A maximum of 10 measurements (5 before and 5 after infusion of a drug) per patient will be performed.
  We want to explicitly mention that for study purposes the surgery or anesthesia will never be prolonged or modified, nor will any drugs be give for study purposes.
  Other Names: epihedrine; nitroprusside; nicardipine

SUMMARY:
Hypertension affects 32-35% of the global adult population. Despite many drugs being available hypertension is not controlled in 50% of the over 500 million treated people leaving patients with an elevated blood pressure for life.

In the development of isolated systolic hypertension, the aorta plays a pivotal role. With each heartbeat, the heart empties its stroke volume into the large arteries. These arteries, particularly the thoracic part of the aorta, temporarily distend to buffer the stroke volume and thereby dampen the pressure fluctuation: they have a Windkessel function. When this function is reduced (and arterial stiffness is increased), the heart needs to contract more forcefully during ejection, leading to isolated systolic hypertension.

Likely, the aorta is not just a passive structure (the aorta as an elastic 'bicycle tube'). Rather, the smooth muscle cells in the aorta wall can presumably actively change the aorta's dimension through vasoconstriction/-dilation. If this is the case, such vasoconstriction/-dilation will have direct consequences for the aorta's Windkessel function and, since this Windkessel function directly influences the blood pressure flucturation, also for hypertension and its progression. Therefore, the aim of this study is to quantify the thoracic aorta's ability to vasoconstrict, and to assess whether this contractility is related to specific predictors.

During the study we will measure in the operating room the thoracic descending and ascending aortic diameter with transoesopahgeal echocardiography (part of standard clinical care), before and after administration of vasoactive drugs (phenylephrine and norepinephrine; also part of standard clinical care). During these measurements we will simultanesouly measure peripheral arterial blood pressure and an electrocardiogram (ECG, to monitor sympathetic activity as estimated using heart rate variability analysis). Measurements will be performed at Catharina Hospital Eindhoven, the Netherlands (NL), where patients undergo elective cardiac surgery. Using the data obtained, we will 1) establish and quantify the in vivo contractility of the human thoracic aorta, and 2) study whether and to which extent potential predictors (age, sex, smoking status, antihypertensive medication use/class, mean arterial pressure, pulse pressure as an indirect measure of arterial stiffness, diabetes, chronic kidney disease, total cholesterol, and sympathetic activity) influence contractility

DETAILED DESCRIPTION:
At the OR, the patient will be sedated and have a transoesophageal echo (TEE) catether inserted, which is part of standard clinical care. When a patient becomes hypotensive and the attending anesthesiologist decides to infuse any of the following drugs (phenylephrine, ephedrine, norepinephrine, nitroprusside, or nicardipine), before infusion, the anesthesiolgist will acquire with TEE 10 beats of the thoracic ascending and descending aorta respectively. This is defined as one measurement. Five minutes after infusion the same measurement is repeated. A maximum of 10 measurements (5 before and 5 after infusion of a drug) per patient will be performed.

The investigators want to explicitly mention that for study purposes the surgery or anesthesia will never be prolonged or modified, nor will any drugs be give for study purposes.

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery

Exclusion Criteria:

* No informed consent for study participation Atrial fibrillation or other cause of irregular heart rhythm Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who undergo elective cardiac surgery
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-05-27 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
To establish and quantify the in vivo contractility of the human thoracic aorta | 1 month
  The primary outcome used in this statistical analysis is the relative contractile isobaric (pressure-normalised) cross-sectional area change of the thoracic aorta (ΔCSA) to phenylephrine (ΔCSAPE).

SECONDARY OUTCOMES:
To quantify the magnitude of contractile response | 2 months
  To quantify the magnitude of contractile response ΔCSAPE with 95% confidence (α=0.05) and ≤2.5% margin of error
To study whether and to which extent potential predictors influence contractility. | 3 months
  to identify predictors of the contractile response and build a realistic statistical model, in addition to using 1) pulse pressure as an indirect measure of arterial stiffness, we will assess the effects of additional potential predictors: age, sex (M/F), smoking status (yes/no), antihypertensive medication use (none/calcium channel blockers/renin-angiotensin system blockers/diuretics/nitrates, mean arterial pressure, diabetes (yes/no), chronic kidney disease (yes/no), total cholesterol, and sympathetic activity. ΔCSAPE will be expressed as a relative (with respect to pre-contraction CSA) value to account for variations in aorta size among patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina hospital, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No
Raw hemodynamic data as the ultrasound acquisitions will be stored on a local server at Catharina Hospital only accessible to members of the study team. Patient characteristics, hemodynamic interventions, and laboratory results will be recorded in an electronic CRF. The CRF does not contain data that can be linked to the patient. Instead of this, a subject identification code is used in the CRF to link data to the patient if needed. The key to the code is safeguarded by the investigators.